CLINICAL TRIAL: NCT05196776
Title: Diagnostic Accuracy of a Portable, Handheld Point-of-Care Ultrasound Device vs a Traditional Cart-Based Model
Brief Title: Diagnostic Accuracy of Handheld vs Traditional Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 28766
Record Dates: First submitted 2021-12-06; First posted 2022-01-19 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Image, Body

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Portable, Handheld Device (Experimental): Patients will receive a point-of-care ultrasound using a handheld, portable ultrasound device.
  Interventions: Device: Portable, handheld point-of-care ultrasound device
- Traditional, Cart-based Ultrasound (Active Comparator): Patients will receive a point-of-care ultrasound using a traditional, cart-based ultrasound machine.
  Interventions: Device: Cart-based point-of-care ultrasound device

INTERVENTIONS:
Device: Portable, handheld point-of-care ultrasound device — The patient will have an ultrasound performed using a handheld, portable device.
  Arms: Portable, Handheld Device
Device: Cart-based point-of-care ultrasound device — The patient will have an ultrasound performed using a traditional cart-based model.
  Arms: Traditional, Cart-based Ultrasound

SUMMARY:
Patients receiving a point-of-care ultrasound will be randomized into a portable, handheld device or a traditional cart-based ultrasound machine to compare diagnostic capability.

DETAILED DESCRIPTION:
Patients who require a point-of-care ultrasound examination of their kidneys, gallbladder, heart, lung, or aorta will be enrolled. Once enrolled, the patient will be randomized to receive the point-of-care ultrasound using a portable, handheld ultrasound or a traditional cart based model. The ultrasound examinations will be performed by emergency medicine post-graduate year 1-3 residents or an ultrasound fellow and reviewed by the supervising emergency medicine attending physicians credentialed in performing and interpreting point-of-care ultrasound.

Based on the clinical presentation, the provider will perform one of the following ultrasounds: cardiac to assess ejection fraction ( <50%, 30-50%, <30%), lung to assess for presence or absence of B-lines, gallbladder to assess for the presence or absence of gallstones, renal to assess for the presence or absence of hydronephrosis, or aorta to assess for the presence or absence of an aneurysm. The diagnostic accuracy of the portable, handheld and the cart-based model will be assessed using the following as the diagnostic standard: cardiology-interpreted echocardiogram, radiology-interpreted ultrasound or computed tomography, or quality review of the point-of-care ultrasound by 3 ultrasound fellowship trained physicians.

ELIGIBILITY:
Inclusion Criteria:

1. English and Spanish-speaking patients, who require a gallbladder, cardiac, renal, aorta, or lung ultrasound based on the discretion of the treating physician.

Exclusion Criteria:

1. All other non-English and non-Spanish speaking patients
2. Vulnerable groups
3. Patients unable to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Portable, Handheld Device | Traditional, Cart-based Ultrasound
Started | 54 | 56
Completed | 53 | 56
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portable, Handheld Device | Traditional, Cart-based Ultrasound | Total
Number analyzed (Participants) | 53 | 56 | 109
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [18 to 89] | 57 [18 to 90] | 59 [18 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 26 | 22 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 56 | 109

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: The primary outcome will be difference in diagnostic accuracy between the two methods (the percent of diagnostic accuracy of the hand-held and the percent of diagnostic accuracy of the cart-based model).
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Portable, Handheld Device | Traditional, Cart-based Ultrasound
Number analyzed (Participants) | 54 | 56
Participants | 53 | 56

2. Secondary Outcome: Image Quality by Expert Review
Description: Using a Likert scale of 1-7 (1 = unable to assess image; 7 = highest quality), ultrasound fellowship-trained providers will assess the image quality of images obtained by each provide in the study.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Portable, Handheld Device | Traditional, Cart-based Ultrasound
Number analyzed (Participants) | 53 | 56
score on a scale | 4 [1 to 7] | 5 [1 to 7]

ADVERSE EVENTS:
Time Frame: 1 day
Description: There is no risk associated with point-of-care ultrasound.
Arm/Group | Portable, Handheld Device | Traditional, Cart-based Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 0/54 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT05196776/Prot_SAP_000.pdf